CLINICAL TRIAL: NCT03686150
Title: Vitamin D Oral Replacement in Asthma
Acronym: VDORA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IDeA States Pediatric Clinical Trials Network (Network)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 101; U24OD024957 (NIH)
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Results first posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-03

CONDITIONS: Asthma; Vitamin D Deficiency; Pediatric Obesity
Keywords: pediatric obesity
MeSH Terms: conditions — Asthma; Vitamin D Deficiency; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, parallel arm clinical trial 4 arms in part 1 2 arms in part 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part 1, Cohort 1 Vitamin D3 oral regimen (Experimental): Intervention: Vitamin D: Single 50,000 IU loading dose + 6000 IU daily dose
  Interventions: Dietary Supplement: Vitamin D3 oral regimen
- Part 1, Cohort 2 Vitamin D3 oral regimen (Experimental): Vitamin D: Single 50,000 IU loading dose + 10,000 IU daily dose
  Interventions: Dietary Supplement: Vitamin D3 oral regimen
- Part 1, Cohort 3 Vitamin D3 oral regimen (Experimental): Vitamin D: 6000 IU daily dose
  Interventions: Dietary Supplement: Vitamin D3 oral regimen
- Part 1, Cohort 4 Vitamin D3 oral regimen (Active Comparator): Vitamin D: 600 IU daily dose
  Interventions: Dietary Supplement: Vitamin D3 oral regimen
- Part 2, Cohort A Vitamin D3 oral regimen (Experimental): Vitamin D: Single 50,000 IU loading dose + 8,000 IU daily doseD
  Interventions: Dietary Supplement: Vitamin D3 oral regimen
- Part 2, Cohort B Vitamin D oral regimen (Active Comparator): Vitamin D: 600 IU daily dose
  Interventions: Dietary Supplement: Vitamin D3 oral regimen

INTERVENTIONS:
Dietary Supplement: Vitamin D3 oral regimen — Vitamin D3 oral regimens supplementation

SUMMARY:
The overall objective of the study is to determine the pharmacokinetics of Vitamin D supplementation in children who have asthma and are overweight or obese.

DETAILED DESCRIPTION:
This study has two parts. In part 1, study participants will be randomized to receive one of four doses of vitamin D supplementation in international units (IU) over at 16-week period: 1) Single 50,000 IU loading dose + 6000 IU daily dose; 2) Single 50,000 IU loading dose + 10,000 IU daily dose: 3) 6000 IU daily dose; or 4) 600 IU daily dose. Based on pharmacokinetic analysis, one of the doses (1-3) will be selected to use in part 2.

In part 2, study participants will be randomized to the dose selected in part 1 or the 600 IU daily dose of vitamin D supplementation to be administered over a 16-week dosing period.

Across both parts, safety of each dose regimen of vitamin D supplementation will be evaluated, and the effectiveness of each dose to achieve a serum level of 25(OH)D greater than or equal to 40 ng/ml will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index greater than or equal to 85% for age and sex
* Physician-diagnosed asthma
* Ongoing relationship with asthma provider responsible for asthma care
* Serum 25(OH) D level 10 ng/ml to less than 30 ng/ml at screening visit based on local laboratory test
* Ability to swallow pills similar in size to the vitamin D preparation to be used
* Signed consent form from parent, legal guardian or caregiver and signed assent from participant (as appropriate)
* Females of childbearing years must not be pregnant, must not be lactating and must agree to practice adequate birth control method
* Child and parent, legal guardian, or caregiver must speak English or Spanish

Exclusion Criteria:

* Known diseases of calcium metabolism or the parathyroid
* History of renal insufficiency or kidney stones
* Known liver failure or history of abnormal liver function tests
* History of Williams syndrome, sarcoidosis, or granulomatous disease
* Active tuberculosis
* Spot urine calcium/creatinine ration greater than 0.37 (calcium and creatinine measured in mg/ml). This can be repeated following adequate hydration
* Clinical evidence of rickets
* Taking supplemental vitamin D greater than equal to 1000 IU per day

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Nemours/Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - University of Louisville, Louisville, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Community Medical Center, Missoula, Montana
  - University of Nebraska Medical Center/Children's Hospital and Medical Center, Omaha, Nebraska
  - Dartmouth Hospital - Manchester, Manchester, New Hampshire
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Children's Hospital OU Medical Center, Oklahoma City, Oklahoma
  - University of South Carolina, Columbia, South Carolina
  - University of Vermont Medical Center, Burlington, Vermont
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to Data and Specimen Hub (DASH) of NICHD
Supporting Information: Study Protocol, ICF
Time Frame: Anticipated date of data upload is September 2023
Access Criteria: per DASH requirements

REFERENCES:
- [Background] O'Sullivan BP, James L, Majure JM, Bickel S, Phan LT, Serrano Gonzalez M, Staples H, Tam-Williams J, Lang J, Snowden J; IDeA States Pediatric Clinical Trials Network. Obesity-related asthma in children: A role for vitamin D. Pediatr Pulmonol. 2021 Feb;56(2):354-361. doi: 10.1002/ppul.25053. Epub 2020 Dec 8. PMID 32930511
- [Derived] Lang JE, Ramirez RG, Balevic S, Bickel S, Hornik CP, Majure JM, Venkatachalam S, Snowden J, O'Sullivan B, James L. Pharmacokinetics of Oral Vitamin D in Children with Obesity and Asthma. Clin Pharmacokinet. 2023 Nov;62(11):1567-1579. doi: 10.1007/s40262-023-01285-9. Epub 2023 Aug 30. PMID 37646988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 166 study participants consented to be screened for the trial; 112 met eligibility criteria and were randomized onto the trial.
  The trial comprised of a Dose Finding part (Part 1) and a Dose Confirming par (Part 2). During Part 1, participants (children) were enrolled and randomized to one of four dose groups at 1:1:1:1 allocation ratio. During Part 2, participants (children) were randomized to one of two dose groups at 2:1 allocation ratio.
Period: Overall Study
Arm/Group | Part 1, Cohort 1 Vitamin D3 Oral Regimen | Part 1, Cohort 2 Vitamin D3 Oral Regimen | Part 1, Cohort 3 Vitamin D3 Oral Regimen | Part 1, Cohort 4 Vitamin D3 Oral Regimen | Part 2, Cohort A Vitamin D3 Oral Regimen | Part 2, Cohort B Vitamin D Oral Regimen
Started | 13 | 12 | 11 | 12 | 43 | 21
Completed | 11 | 10 | 10 | 12 | 42 | 18
Not Completed | 2 | 2 | 1 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 1 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This vitamin D supplementation study was performed in two parts: 1) PK analysis to identify recommended dost for part 2, and 2) assess the effectiveness of the recommended 16-week dosing regimen to achieve serum level of 25(OH)D greater than or equal to 40 ng/mL.
Groups:
- Part 2, Cohort A Vitamin D3 Oral Regimen: Vitamin D: Single 50,000 IU loading dose + 8,000 IU daily dose
  Vitamin D3 oral regimen: Vitamin D3 oral regimens supplementation
- Total: Total of all reporting groups
Arm/Group | Part 1, Cohort 1 Vitamin D3 Oral Regimen | Part 1, Cohort 2 Vitamin D3 Oral Regimen | Part 1, Cohort 3 Vitamin D3 Oral Regimen | Part 1, Cohort 4 Vitamin D3 Oral Regimen | Part 2, Cohort A Vitamin D3 Oral Regimen | Part 2, Cohort B Vitamin D Oral Regimen | Total
Number analyzed (Participants) | 13 | 12 | 11 | 12 | 43 | 21 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (3.1) | 12.3 (3.4) | 11.5 (3.6) | 12.5 (2.9) | 12.2 (2.5) | 11.7 (2.6) | 12.1 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 5 | 5 | 20 | 10 | 53
  Male | 7 | 5 | 6 | 7 | 23 | 11 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 2 | 1 | 7 | 3 | 20
  Not Hispanic or Latino | 7 | 10 | 8 | 10 | 33 | 18 | 86
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 3 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 3 | 1 | 4
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 6 | 4 | 5 | 6 | 15 | 9 | 45
  White | 4 | 5 | 3 | 5 | 19 | 10 | 46
  More than one race | 0 | 1 | 1 | 1 | 2 | 1 | 6
  Unknown or Not Reported | 3 | 1 | 1 | 0 | 3 | 0 | 8
Baseline Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.9 (8.4) | 29.7 (6.4) | 30.1 (4.3) | 32.2 (9.2) | 30.8 (6.9) | 30.3 (8.2) | 31.0 (7.3)
BMI percentile [Count of Participants; unit: Participants]
  >= 85th to < 95th | 3 | 2 | 2 | 3 | 9 | 5 | 24
  >= 95th to < 99th | 4 | 3 | 2 | 3 | 16 | 8 | 36
  >= 99th | 6 | 7 | 7 | 6 | 18 | 8 | 52
Rural-Urban Commuting Area (RUCA) codes [Count of Participants; unit: Participants] — The RUCA codes classify US census tract based on measures of urbanization, population density, and daily commuting from the decennial census. The classification contains whole numbers (1-10) used to delineate metropolitan (1-3), micropolitan (4-6), small town (7-9), and rural areas (10).
  Participants
    Metropolitan | 13 | 10 | 9 | 11 | 32 | 17 | 92
    Micropolitan | 0 | 1 | 1 | 0 | 5 | 1 | 8
    Small town | 0 | 1 | 1 | 1 | 3 | 2 | 8
    Rural | 0 | 0 | 0 | 0 | 3 | 1 | 4
Baseline 25(OH)D [Mean (Standard Deviation); unit: ng/mL] — 25(OH)D = (25-hydroxy vitamin D); Baseline measures were captured at visit 2 (day 0; week 1). Population: Note: Cohort 1, Cohort A, and Cohort B each one participant with missing 25(OH)D measurement at baseline.
  ng/mL
    number analyzed (Participants) | 12 | 12 | 11 | 12 | 42 | 20 | 109
    (all) | 18.3 (6.5) | 20.8 (7.2) | 19.0 (5.2) | 17.6 (5.8) | 17.7 (6.0) | 16.3 (5.2) | 18.0 (6.0)
Baseline 25(OH)D level > 100 ng/mL [Count of Participants; unit: Participants] — 25(OH)D = (25-hydroxy vitamin D) Population: Note: Cohort 1, Cohort A, and Cohort B each had one participant with missing 25(OH) D values at baseline.
  Participants
    number analyzed (Participants) | 12 | 12 | 11 | 12 | 42 | 20 | 109
    Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0
    No | 12 | 12 | 11 | 12 | 42 | 20 | 109

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Optimal Dosing Level to Use in Part 2
Description: Determine the best vitamin D supplementation level based on PK analysis of participants enrolled in Part 1. The PK of 25(OH)D after vitamin D supplementation in children will be characterized using a 2-compartment population PK model (popPK) with linear absorption and elimination kinetics.
Time Frame: 20 weeks
Population: A total of 263 PK samples from 48 participants were collected in part 1 of the VDORA1 study. For the population PK analysis, 36 samples with missing prior dosing information from 13 participants were excluded, leaving a final analysis population of 44 participants with 227 serum concentrations.
Measure: Number; unit: IU
Units Other Than Participants: Serum Concentrations
Groups:
- Vitamin D3 Oral Regimen: Vitamin D: Single 50,000 IU loading dose + 8,000 IU daily dose
  Vitamin D3 oral regimen: Vitamin D3 oral regimens supplementation
Arm/Group | Vitamin D3 Oral Regimen
Number analyzed (Participants) | 44
Number analyzed (Serum Concentrations) | 227
IU
  Daily Dose (IU) | 8000
  Single Loading Dose (IU) | 50000
Statistical Analysis 1: Comparison: Vitamin D3 Oral Regimen; Part 1 of this study was to perform a population PK analysis of 25(OH)D after oral administration of Vitamin D in children who are overweight or obese and have asthma. Based on the interim analysis of the VDORA study, the PK of 25(OH)D after Vitamin D supplementation in children was well characterized by a 2-compartment population PK model with linear absorption and elimination kinetics. A loading dose of 50,000 IU followed by a daily dose of 8,000 IU was recommended; Test type: Other — This was a population PK analysis of 25(OH)D after oral administration of Vitamin D; Based on the interim analysis of the VDORA study, the PK of 25(OH)D after Vitamin D supplementation in children was well characterized by a 2-compartment population PK model with linear absorption and elimination kinetics. A loading dose of 50,000 IU followed by a daily dose of 8,000 IU was recommended

2. Primary Outcome: Part 2: Proportion of Participants With Vitamin D Levels >= 40 ng/ml
Description: Proportion of participants in part 2 who achieve vitamin levels >= 40 ng/ml
Time Frame: 16 weeks
Population: One participant from Cohort A and three participants from Cohort B did not have 25(OH)D measurements at Visit 6 (week 16).
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Part 2, Cohort A Vitamin D3 Oral Regimen | Part 2, Cohort B Vitamin D Oral Regimen
Number analyzed (Participants) | 42 | 18
proportion of participants | 0.786 [0.641 to 0.883] | 0 [0 to 0.176]
Statistical Analysis 1: Comparison: Part 2, Cohort A Vitamin D3 Oral Regimen; This is a one-sample test of proportion; Test type: Other — This is one-sample test of proportion testing the null hypothesis that the proportion of participants with 25(OH)D level >= 40 ng/mL is 50%; p = 0.0001, z-test

ADVERSE EVENTS:
Time Frame: Participant Duration: 30 weeks (2-week screening/run-in; 16-week intervention; 12-week follow-up period)
Description: Using standard definitions of adverse events, adverse events were reported during the intervention and follow-up periods.
Arm/Group | Part 1, Cohort 1 Vitamin D3 Oral Regimen | Part 1, Cohort 2 Vitamin D3 Oral Regimen | Part 1, Cohort 3 Vitamin D3 Oral Regimen | Part 1, Cohort 4 Vitamin D3 Oral Regimen | Part 2, Cohort A Vitamin D3 Oral Regimen | Part 2, Cohort B Vitamin D Oral Regimen
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/11 | 0/12 | 0/43 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/12 | 1/11 | 1/12 | 0/43 | 1/21
Other Adverse Events (participants affected / at risk) | 11/13 | 9/12 | 11/11 | 10/12 | 21/43 | 14/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, Cohort 1 Vitamin D3 Oral Regimen (N=13) | Part 1, Cohort 2 Vitamin D3 Oral Regimen (N=12) | Part 1, Cohort 3 Vitamin D3 Oral Regimen (N=11) | Part 1, Cohort 4 Vitamin D3 Oral Regimen (N=12) | Part 2, Cohort A Vitamin D3 Oral Regimen (N=43) | Part 2, Cohort B Vitamin D Oral Regimen (N=21)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 — In all cases, this SAE was not related to Vitamin D or study procedure.
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 — This SAE was not related to Vitamin D or study procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, Cohort 1 Vitamin D3 Oral Regimen (N=13) | Part 1, Cohort 2 Vitamin D3 Oral Regimen (N=12) | Part 1, Cohort 3 Vitamin D3 Oral Regimen (N=11) | Part 1, Cohort 4 Vitamin D3 Oral Regimen (N=12) | Part 2, Cohort A Vitamin D3 Oral Regimen (N=43) | Part 2, Cohort B Vitamin D Oral Regimen (N=21)
abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
acarodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
adenoidectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
adenotonsillectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
amebiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
asthma (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 2
asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 5 | 3 | 1 | 3
cardiac ablation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
chest cold (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 1
contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 5 | 3 | 2 | 2
depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
diarrhea (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0
dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
ear infection (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 0
ear injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0
emotional disorder of childhood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
eosinophilic oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
epixtaxis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
eyelid sensory disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
fatigue (General disorders) | 1 | 0 | 1 | 0 | 1 | 0
fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
gastritis viral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
gastroenteritis viral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
gastrointestinal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
headache (Nervous system disorders) | 0 | 3 | 3 | 2 | 3 | 1
hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 3
influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
influenza b virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
insomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0
lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 1 | 1 | 1
nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 2
nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
ocular discomfort (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
oropharyngeal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 1 | 1
pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
paresthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
peripheral coldness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
pharyngitis streptococcal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
polydipsia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
post procedural discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
procedural pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
pyrexia (General disorders) | 0 | 0 | 0 | 3 | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 1 | 2 | 0
respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
respiratory tract infection viral (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
scar excision (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
seasonal allergy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
thermal burning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
tinea pedis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
tonsillectomy (Surgical and medical procedures) | 0 | 0 | 1 | 1 | 0 | 0
tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
turbinectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
turbinoplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
upper respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 1
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1 | 0
urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
urine calcium/creatinine ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
vessel puncture site bruise (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
vessel puncture site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0 | 0
vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 1 | 1
wisdom teeth removal (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT03686150/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT03686150/ICF_000.pdf